CLINICAL TRIAL: NCT07014813
Title: Mini Open Subpectoral Press Fit Biceps Tenodesis
Brief Title: Mini-Open Subpectoral Biceps Tenodesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Abd ElGhafour Abd ElRady, Assistant Lecturer at Department of Trauma and orthopedics, Faculty of Medicine, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-1910-2024
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Bicep Tendinitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Candidate Group (Other): The Candidate Group Patients were 30 patients:
  * Seventeen females and Thirteen males with a mean age of 44.4 years (range: 30-60 years).
  * Eight patients were smokers, and ten suffered from controlled diabetes.
  * Three patients were suffering from isolated biceps tendinopathy without associated pathology, Nine were suffering from frozen shoulder, Fifteen patients with different degrees of rotator cuff tears, and the last three patients had biceps slap lesions which were irreparable with anchors.
  * There were 21 dominant and 9 non-dominant shoulders.
  Interventions: Procedure: Sub pectoral fixation

INTERVENTIONS:
Procedure: Sub pectoral fixation — Subpectoral biceps tenodesis via mini-open incision. Biceps tendon prepared with Krackow sutures, press-fit into bony tunnel using harvested bone plug. Stability checked post-fixation.

SUMMARY:
Surgical management of long head of biceps (LHB) lesions is frequent, often alongside other shoulder issues. When conservative treatment fails, tenotomy (for low-demand patients) or tenodesis (preferred for active individuals) is performed. Subpectoral tenodesis offers advantages, and this study assesses a novel press-fit bony plug technique for this approach, evaluating its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Biceps tendon pathologies after failure of conservative measures: biceps tenosynovitis, recurrent subluxation, or SLAP lesions.
* Young and middle-aged individuals (20-60 years old).

Exclusion Criteria:

* Patients with avascular necrosis or arthritis.
* Extensive bone loss.
* Poor bone density.
* Active infection.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients reported having at least a 50% Increase in their Amircan Shoulder and Elbow Society (ASES) Scoring, and decrease in their pain (measured according to VAS score) with no loss in the range of motion. | 42 Months
  The Success rate of sub-pectoral fixation of the biceps tendon was assessed as that there was proportion of patients who achieved a clinically significant improvement in shoulder and elbow function (at least a 50% increase in ASES score), a notable reduction in pain (decrease in VAS score), while maintaining their ange of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Kasr Al-Einy, Cairo, Egypt